CLINICAL TRIAL: NCT04301180
Title: Effectiveness of a Multicompetent Intervention on the Quality of the Diet in the Preschool Population
Brief Title: Quality of Diet in Preschool Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Collaborators: David Varillas Delgado (Unknown); María Cristina Martincrespo-Blanco (Unknown); Saray Blanco-Abril (Unknown); María Gema Cid-Expósito (Unknown); Juana Robledo-Martín (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEIC 2016/013
Record Dates: First submitted 2020-02-29; First posted 2020-03-10 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-08

CONDITIONS: Feeding and Eating Disorders of Childhood
Keywords: Nutritional Status; Child Nutrition Sciences; Nutrition Therapy; Nutrition Assessment; Diet, Food, and Nutrition
MeSH Terms: conditions — Feeding and Eating Disorders of Childhood

STUDY DESIGN:
Intervention Model Description: The experimental group conducted 10 weekly sessions, with an approximate duration of 45 minutes per session, which consisted of the presentation of food education content while conducting an orchard with seasonal vegetables. Simple recipes were also described in which these vegetables were included to be made at home, along with information from children's books that dealt with the topic of food and were available in the public library.
  The control group received the usual training corresponding to the contents of the "human body" module that is currently taught in each center.
  All children in the experimental groups were given written instructions so that they could perform at their home, together with their parents, the manipulative activities suggested each week. All these contents were common for all the participants in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The experimental group conducted 10 weekly sessions, with an approximate duration of 45 minutes per session, which consisted of the presentation of food education content while conducting an orchard with seasonal vegetables. Simple recipes were also described in which these vegetables were included to be made at home, along with information on children's books that dealt with the topic of food and were available in the public library.
  All children in the experimental groups were given written instructions so that they could perform at their home, together with their parents, the manipulative activities suggested each week. All these contents were common for all the participants in the study. Session material was renewed weekly.
  Interventions: Device: Education food
- Control (No Intervention): The control group received the usual training corresponding to the contents of the "human body" module that is currently taught in each center.

INTERVENTIONS:
Device: Education food — The intervention consisted of the presentation of food education content while conducting an orchard with seasonal vegetables
  Arms: Experimental

SUMMARY:
Childhood obesity is a problem of high prevalence and repercussions in adulthood. It is mostly due to inadequate life habits, modifiable through preventive strategies. The objective was to evaluate in the medium term the effectiveness of an intervention on adherence to the Mediterranean diet pattern in preschoolers.

Method: Community trial with two groups, in children between 3-5 years. The experimental group conducted a school garden and the usual contents on human body and health were taught in the control. Two schools were selected by cluster sampling, whose first unit of randomization were the educational areas followed by schools. The adaptation to the Mediterranean diet pattern was evaluated using the KIDMED questionnaire and weight, height, BMI and sociodemographic variables were controlled.

ELIGIBILITY:
Inclusion Criteria:

* Age between 3 and 5 years
* Oral comprehension of Spanish.

Exclusion Criteria:

* Existence of language barriers in parents defined as not understanding spoken or written Spanish.
* Treatment with glucocorticoids.
* Having chronic diseases that could interfere with somatometry.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Change of KIDMED questionnaire | During the procedure; baseline, 1 year and 2 years
  Mediterranean diet adherence assessment questionnaire, 16 items, scored of 1 point per item, minimun 0 points (worse) to 16 points (better).

SECONDARY OUTCOMES:
Change of Weight | During the procedure; baseline, 1 year and 2 years
  Changes of Weight in kilograms (Kg), were collected in children using approved scale at baseline, al 1 year and 2 years.
Educational level of parents | Baseline
  A survey will assess the level of education of parents; primary, secondary, university or without education, expressed in %.
Employment status of parents | Baseline
  The parents' purchasing level will be evaluated in percentages (%); low, medium and high employement status.
Change of Height | During the procedure; baseline, 1 year and 2 years
  Changes of Height in meters, were collected in children using approved scale at baseline, al 1 year and 2 years.
Change of BMI (body mass index) | During the procedure; baseline, 1 year and 2 years
  Change of weight and height outcomes will be combined to report BMI in kg/m^2, upper 20 is considered obesity.

CONTACTS AND LOCATIONS:
Locations (1):
- David Varillas Delgado, Pozuelo de Alarcón, Madrid, Spain